CLINICAL TRIAL: NCT02529098
Title: Modification in Cortical Activation by Functional Magnetic Resonance Imaging (fMRI) in Pseudophakic Patients With Visual Difficulties After a Multifocal Implantation
Brief Title: Modification in Cortical Activation in Pseudophakic Patients With Visual Difficulties After a Multifocal Implantation
Acronym: PlainteIMF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: default recruitment
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 12 523 03
Record Dates: First submitted 2015-06-10; First posted 2015-08-19 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Vision Disorders
Keywords: functional magnetic resonance imaging; Lens implantation; pseudophakia
MeSH Terms: conditions — Vision Disorders; Pseudophakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- asymptomatic patients (Sham Comparator): fMRI Asymptomatic patients
  Interventions: Other: fMRI
- symptomatic patients (Experimental): fMRI patients with visual difficulties
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — functional magnetic resonance imaging

SUMMARY:
This study will highlight differences in cortical activation between asymptomatic and symptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Cataract surgery with an bilateral multifocal lens implant Restor

Symptomatic patients :

* Symptomatic bilateral visual difficulties for 3 months or more after the intervention which impact the daily activity

Asymptomatic patients :

* No visual complaint for 3 months or more after the intervention

Exclusion Criteria:

* Patients with ophthalmology disorders
* Contra indication for fMRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Extent of neural activation in visual cortex measured by the number of voxels | 1 day
  compare the extent of neural activation in visual cortex between groups

SECONDARY OUTCOMES:
extent of neural activation in visual cortex measured by the number of voxels | 1 day
  compare the extent of neural activation in the different area visual cortex between groups

CONTACTS AND LOCATIONS:
Overall Officials: Francois Malecaze, professor, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France